CLINICAL TRIAL: NCT00699569
Title: The Effect of Hyperimmune Colostrum on Radiation-Induce Oral Mucositis of Patients With Head and Neck Cancer
Brief Title: Hyperimmune Colostrum and Oral Mucositis
Acronym: Mucositis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Nachum Vaisman Prof', Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: TASMC-08-NV-248; 0248-08-TLV
Record Dates: First submitted 2008-06-17; First posted 2008-06-18 (Estimated); Last update posted 2008-07-23 (Estimated); Status verified 2008-06

CONDITIONS: Head and Neck Cancer
Keywords: hyperimmune colostrum; mucositis
MeSH Terms: conditions — Head and Neck Neoplasms; Mucositis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Patients receiving active investigational product
  Interventions: Dietary Supplement: hyperimmune colostrum
- 2 (Placebo Comparator): Patients receiving Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: hyperimmune colostrum — hyperimmune colostrum
  Arms: 1
Dietary Supplement: Placebo
  Arms: 2

SUMMARY:
To study the effect of daily intake of hyperimmune colostrum on prevention and treatment of oral mucositis in patients with head and neck cancer undergoing high-dose radiation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with: naso-pharynx, oral cavity, oro-pharynx and advanced localized laryngeal cancer.

Exclusion Criteria:

* Other tumors
* Non-epithelial tumors
* Pregnancy
* Poor functional status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-07 (Estimated); Study Completion 2009-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Nachum Vaisman, Prof', Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Sourasky Medical Center, Tel Aviv, Israel